CLINICAL TRIAL: NCT00747045
Title: A Prospective Single Blind Controlled Study to Assess the Efficacy of a Lung Protective Ventilation Strategy in the Prevention of Reperfusion Lung Injury Following PTE
Brief Title: Lung Protective Ventilation in Pulmonary Thromboendarterectomy (PTE) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Kim Kerr, Clinical Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 080721
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension; Acute Lung Injury
Keywords: Chronic Thromboembolic Pulmonary Hypertension; Lung Injury; Ventilation Strategies
MeSH Terms: conditions — Acute Lung Injury; Lung Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low tidal volume (Experimental): Tidal volume of 6 mL/Kg ideal body weight
  Interventions: Other: Ventilation Strategy
- Usual care (Active Comparator): Tidal volume of 10 mL/Kg ideal body weight
  Interventions: Other: Ventilation Strategy

INTERVENTIONS:
Other: Ventilation Strategy — Comparison of low vs standard tidal volumes in patients undergoing PTE

SUMMARY:
Chronic thromboembolic pulmonary hypertension (CTEPH) is caused by unresolved thromboemboli in the pulmonary arteries, which lead to pulmonary hypertension and, left untreated, right heart failure. This disease can be potentially cured by performing a pulmonary thromboendarterectomy (PTE) to remove the blood clots. The surgery is not without risk and the most worrisome complication is the development of a form of acute lung injury called reperfusion lung injury, which occurs in about 40 percent of patients.

The landmark publication of the ARDSNET study demonstrated that a low tidal volume strategy of mechanical ventilation, decreased morbidity and mortality in patients who had acute respiratory distress syndrome (ARDS). Since then there have been some studies examining the role of a low tidal volume strategy in all patients who are mechanically ventilated. Some studies have demonstrated a decreased incidence of acute lung injury while others have failed to do the same. In patients at high risk for developing acute lung injury, such as patients undergoing PTE, there may be a benefit to using low tidal volumes to reduce the incidence of reperfusion lung injury.

To assess the efficacy of a low tidal volume ventilation strategy in patients undergoing PTE, 134 patients will be randomized at the time of surgery to either low tidal volumes (6ml/kg of ideal body weight), or standard tidal volumes (10ml/kg of ideal body weight). Patients will be followed clinically to assess for the development of reperfusion lung injury. This will be defined as the development of hypoxemia (PaO2/FiO2 ratio less than 300) and chest infiltrates in the area of reperfused lung with no other identifiable etiology within the first 72 hours of surgery. Patients will also be assessed for other factors known to contribute to acute lung injury including: plateau pressures, peak inspiratory pressures, fluid balance, and number of transfusions received. Secondary endpoints of the study will be: time to successful spontaneous breathing trial, ventilator free days, ICU free days, hospital free days, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age
* Evidence of CTEPH
* Acceptable surgical candidate

Exclusion Criteria:

* BMI > 40
* Patient undergoing lung biopsy or CABG at time of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2008-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Reperfusion Lung Injury | 72 Hours

SECONDARY OUTCOMES:
ICU free days | 28 days
Hospital Free Days | 28 days
Mortality | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Kim M Kerr, MD, Principal Investigator — UCSD Medical Center
Locations (1):
- UCSD - Thornton Hospital, La Jolla, California, United States

REFERENCES:
- [Derived] Bates DM, Fernandes TM, Duwe BV, King BO, Banks DA, Test VJ, Fedullo PF, Kim NH, Madani MM, Jamieson SW, Auger WR, Kerr KM. Efficacy of a Low-Tidal Volume Ventilation Strategy to Prevent Reperfusion Lung Injury after Pulmonary Thromboendarterectomy. Ann Am Thorac Soc. 2015 Oct;12(10):1520-7. doi: 10.1513/AnnalsATS.201503-142OC. PMID 26241077